CLINICAL TRIAL: NCT00762905
Title: A Prospective, Randomised, Controlled, Double-masked, Multi-center Clinical Trial of MedLogic LiquiBand Laparoscopic Versus Dermabond in the Closure of Surgical Incisions
Brief Title: Clinical Trial of MedLogic LiquiBand Laparoscopic Versus Dermabond in the Closure of Surgical Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedLogic Global Limited (Industry)
Responsible Party: Richard Stenton, MedLogic Global Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDL-0601
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Laparoscopic Surgery
Keywords: cyanoacrylate; LiquiBand Laparoscopic; Dermabond; The rate of complete dermal apposition; The rate of wound infections and wound dehiscence; The rate of optimal cosmesis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): LiquiBand Laparoscopic
  Interventions: Device: LiquiBand Laparoscopic
- 2 (Active Comparator): Dermabond
  Interventions: Device: Dermabond

INTERVENTIONS:
Device: LiquiBand Laparoscopic — LiquiBand Laparoscopic™ is a sterile, liquid adhesive made up of a blend of n-butyl and 2-octyl cyanoacrylate intended for soft tissue approximation of skin wounds. It is packaged in a sterile, single-use, nylon applicator with internal glass ampoule containing 0.8g of adhesive and sealed in a PETG/Tyvek blister pack. LiquiBand Laparoscopic™ is intended to be applied topically to pre-apposed wound edges. The tissue adhesive sets rapidly (5 - 10 seconds) to hold the wound closed. Following wound closure the product is designed to apply a broad coverage of adhesive to act as a liquid dressing to protect the wound.
  Arms: 1
Device: Dermabond — High viscosity DermaBond Topical Skin Adhesive is a sterile, liquid topical skin adhesive containing a monomeric (2-octyl cyanoacrylate) formulation and the colorant D & C Violet #2. It is provided in a single use applicator packaged in a blister pouch. The applicator is comprised of a crushable glass ampule contained within a plastic vial with attached applicator tip. As applied to skin, the liquid is syrup-like in viscosity and polymerizes within minutes.
  Arms: 2

SUMMARY:
To evaluate the effectiveness, safety, and utility of LiquiBand Laparoscopic™ in relation to a currently approved active control product (High Viscosity DermaBond). Specifically, the study is powered to demonstrate that LiquiBand Laparoscopic™ is not inferior to DermaBond in the rates of infection, dehiscence, cosmesis and apposition of the skin.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, double-masked multi-center clinical trial. Patients requiring laparoscopic surgery will be enrolled and randomized to receive either LiquiBand Laparoscopic™ or DermaBond High Viscosity for incision closure. No other closure methods will be allowed. All eligible laparoscopic incisions per patient will be enrolled. Patients will be followed at 2 weeks and 3 months post-procedure to assess wound characteristics, wound infection, wound dehiscence and at 3 months for cosmesis. The study will be double-masked in that both the wound evaluator and patient will be masked to the randomized study treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a laparoscopic surgical procedure
* Aged 18 years or older
* Agree to return to 2-weeks (3 days) post-procedure follow-up visit
* Agree to return to 3-month (5 days) post-procedure follow-up visit
* Able and willing to give informed consent and to comply with all study requirements

Exclusion Criteria:

* Known sensitivity to cyanoacrylate, formaldehyde or acetone products,
* Surgical procedures involving mucus membranes or eyes
* History of skin rashes or exfoliative condition at time of procedure
* History of keloid formation or hypertrophy
* Currently on immunosuppressive therapy
* Decubitus ulcer
* Pregnant or nursing.
* Participated in an investigational drug or device study within the past 3 months
* Conditions known to interfere with wound healing:
* Diabetes, Type I or II
* Advanced chronic renal insufficiency (GFR greater than 25 mL/min or with clinical signs of azotemia), uremia or endstage renal disease
* Advanced liver failure or cirrhosis (Child-Pugh score of B or C)
* Advanced malignancy, or cancer patients currently receiving chemotherapy (within 30 days of procedure)
* History of radiation therapy to the study area
* Advanced COPD (FEV greater than 1 litre and or PaO2 60 mmHg)
* Suspected infection at incision site
* Peripheral vascular disease
* Corticosteroid therapy
* Morbid obesity (50-100 percent or 100 pounds above their ideal body weight and/or a BMI value greater than 40)
* Blood clotting disorders (e.g. Haemophilia)
* Wounds under high tension forces (over joints)
* Life expectancy of greater than 3 months
* ASA level of 4 or 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The rate of complete dermal apposition at 2-weeks (3 days) To compare the rates of wound infections and wound dehiscence The rate of optimal cosmesis (score=6) at 3-months (± 5 days) will be calculated | 8 to 10 months

SECONDARY OUTCOMES:
Time to close incision Patient and user satisfaction | 8 to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stenton, Study Director — Sponsor Name Pending
Locations (4):
- United Kingdom (4):
  - Milton Keynes General Hospital, Milton Keynes, Bucks
  - Royal Devon and Exeter Hospital (Wonford, Exeter, Devon
  - Royal Surrey County Hospital, Guildford, Surrey
  - Huddesfield Royal Infirmary, Huddersfield, West Yorkshire

REFERENCES:
- [Derived] Kent A, Liversedge N, Dobbins B, McWhinnie D, Jan H. A prospective, randomized, controlled, double-masked, multi-center clinical trial of medical adhesives for the closure of laparoscopic incisions. J Minim Invasive Gynecol. 2014 Mar-Apr;21(2):252-8. doi: 10.1016/j.jmig.2013.10.003. Epub 2013 Oct 12. PMID 24128996